CLINICAL TRIAL: NCT06627673
Title: MultiCenter Prospective Parallel Registry Controlled Investigational Device Exemption Clinical Study to Determine Non-Inferiority of the PEEK-OPTIMA™ Femoral Component Versus a CoCr Alloy Femoral Component of Similar Design for TKA
Brief Title: MultiCenter IDE Study of the PEEK-OPTIMA™ Femoral Component vs a CoCr Alloy TKA Femoral Component of Similar Design
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maxx Orthopedics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PK-00001
Record Dates: First submitted 2024-10-03; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Knee Osteoarthritis
Keywords: Total Knee Replacement; Total Knee Arthroplasty; Polyether-ether-ketone
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Intervention Model Description: This study is a single arm, multi-center, prospective IDE trial. Two hundred (200) patients recruited and consented will receive the PEEK-OPTIMA™ Femoral Component and results will be compared to matched historic controls from the Maxx Orthopedics Freedom Total Knee System product registry (PK-00002 REV-01, WCG IRB# 20241890). Male and female patients 18 years of age or older with Knee Society Score (KSS) of >25 and <75 will be eligible for enrollment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Treatment arm utilizing primary TKA with PEEK femoral component (Experimental): This study is a single arm, multi-center, prospective IDE trial. Two hundred (200) patients recruited and consented will receive the PEEK-OPTIMA™ Femoral Component and results will be compared to matched historic controls from the Maxx Orthopedics Freedom Total Knee System product registry (PK-00002 REV-01, WCG IRB# 20241890). Male and female patients 18 years of age or older with Knee Society Score (KSS) of >25 and <75 will be eligible for enrollment.
  Interventions: Device: Total Knee Arthroplasty

INTERVENTIONS:
Device: Total Knee Arthroplasty — Primary Total Knee Arthroplasty with a PEEK femoral component
  Other Names: Total Knee Replacement

SUMMARY:
The purpose of this investigational device exemption (IDE) study is to monitor the performance (safety and efficacy) of the Maxx Orthopedics, Freedom Total Knee® System, with a femoral component of similar design, manufactured from polyether-ether-ketone (PEEK).

DETAILED DESCRIPTION:
The purpose of this investigational device exemption (IDE) study is to monitor the performance (safety and efficacy) of the Maxx Orthopedics, Freedom Total Knee® System, with a femoral component of similar design, manufactured from polyether-ether-ketone (PEEK).

PEEK is a high-performance, engineering thermoplastic characterized by an unusual combination of properties. These properties range from high temperature performance to mechanical strength and excellent chemical resistance.

The PEEK-OPTIMA® femoral component, is an investigational device and is the subject of this study approved for IDE by the Federal Food and Drug Administration (FDA).

Maxx Orthopedics, Freedom Total Knee System is used with instrumentation to assist with surgery of the knee. The Maxx Orthopedics, Freedom Total Knee System implants are approved by the FDA for use in the United States and is not investigational.

All patients will receive the Freedom Total Knee System with the PEEK femoral component. Patient / study participents' records will be reviewed for identification of any and all complications, post-operative care, component safety and efficacy, and if re-operation is needed.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18 years of age or older.
* Subjects with a primary diagnosis of end-stage symptomatic unilateral primary knee osteoarthritis.
* Subjects with a pre-operative Knee Society Score (KSS) Knee score of >25 and <75.
* Subjects who, in the opinion of the Investigator, can understand this clinical investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups.
* Subjects who can give voluntary, written informed consent to participate in this clinical investigation and from whom consent has been obtained.

Exclusion Criteria:

* Subjects who, in the opinion of the Investigator, have an existing condition that would compromise their participation and follow-up in this clinical investigation.
* Subjects who are known drug or alcohol abusers or with psychological disorders that could affect follow-up care or treatment outcomes.
* Subjects who have participated in a clinical study with an investigational product in the last 6 months.
* Subjects with other significant disabling problems from the muscular-skeletal system other than in the knees (i.e.: muscular dystrophy, polio, neuropathic joints).
* Subjects with known osteoporosis and/or previous history of fracture related to osteoporosis.
* Subjects with a current or active history of malignancy, active or suspected infection, Paget's disease, renal osteodystrophy, immunologically suppressed, rheumatoid arthritis, sickle cell anemia, and systemic lupus erythematosus.
* Subjects defined by the Investigator as American Society of Anesthesiologists (ASA) Grade III or IV.
* Subjects who have a neuromuscular or neurosensory deficit.
* Female subjects who are pregnant or lactating.
* Subjects with an anatomical limb alignment of above 20 degrees varus or valgus.
* Subjects with primary or secondary diagnosis of inflammatory or traumatic arthritis.
* Subjects with a fixed flexion deformity of over 20 degrees.
* Subjects with recurvatum (definition: hyperextension ≥ 5 degrees).
* Subjects who have previously undergone surgery on the indicated knee including total knee arthroplasty, patellofemoral arthroplasty, or unicondylar knee arthroplasty, high tibial osteotomy, ligament reconstruction, fusion, open reduction and internal fixation.
* Subjects that have undergone, or scheduled to undergo, contralateral total knee arthroplasty or unicondylar knee arthroplasty within ±1 year from the study surgical procedure.
* Evidence of active or suspected (systemic or local) infection at time of surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Original Knee Society Score | 24 months post-treatment.
  The Knee Society Score rating system was first introduced during the late 1980's and has become the standard clinical evaluation system for reporting results for patients undergoing Total Knee Arthroplasty. Most major journals strongly encourage that total knee manuscripts include Knee Society Score rating scores as part of the result section. The Knee Society Score consists of points given for pain, range of motion, and stability. The Function Score consists of points given for the ability to walk on level surfaces, and the ability to ascend and descend stairs, with deductions for the use of external supporting devices.
  The Knee Society Score is usually reported as the two scores, "Knee Score" and "Function Score," rather than a summation score. The KSS score has a maximum of 100 points for each domain (Knee and Function).

SECONDARY OUTCOMES:
Knee Society Score (Knee Scores) | Subject reported outcomes at 3-6 weeks 3-, 6-, 12- and 24-months post-treatment
  The Knee Society Score rating system was first introduced during the late 1980's and has become the standard clinical evaluation system for reporting results for patients undergoing Total Knee Arthroplasty. Most major journals strongly encourage that total knee manuscripts include Knee Society Score rating scores as part of the result section. The Knee Society Score consists of points given for pain, range of motion, and stability. The Function Score consists of points given for the ability to walk on level surfaces, and the ability to ascend and descend stairs, with deductions for the use of external supporting devices.
  The Knee Society Score is usually reported as the two scores, "Knee Score" and "Function Score," rather than a summation score. The KSS score has a maximum of 100 points for each domain (Knee and Function).
Knee Society Score (Function Scores) | Subject reported outcomes at 3-6 weeks 3-, 6-, 12- and 24-months post-treatment
  The Knee Society Score rating system was first introduced during the late 1980's and has become the standard clinical evaluation system for reporting results for patients undergoing Total Knee Arthroplasty. Most major journals strongly encourage that total knee manuscripts include Knee Society Score rating scores as part of the result section. The Knee Society Score consists of points given for pain, range of motion, and stability. The Function Score consists of points given for the ability to walk on level surfaces, and the ability to ascend and descend stairs, with deductions for the use of external supporting devices.
  The Knee Society Score is usually reported as the two scores, "Knee Score" and "Function Score," rather than a summation score. The KSS score has a maximum of 100 points for each domain (Knee and Function).
Knee Injury and Osteoarthritis Outcome Score - Joint Replacement (KOOS-JR) | • Subject reported outcomes at 3-6 weeks 3-, 6-, 12- and 24-months post-treatment
  The KOOS-JR is self-administered and assesses three domains: stiffness (1 question), pain (4 questions), function / daily living (2 questions). The KOOS-JR meets basic criteria of outcome measures and can be used to evaluate the course of knee injury and treatment outcome. Each item (questions) is coded from 0 to 4. The raw responses are summed (0-28) which is then converted to an interval score based on the KOOS-JR conversion table. The score is a percentage score from 0 to 100, 0 representing total knee disability and 100 representing perfect knee health.
The Patient Reported Outcomes Measurement Information System (PROMIS) Global-10 | • Subject reported outcomes at 3-6 weeks 3-, 6-, 12- and 24-months post-treatment
  The Patient Reported Outcomes Measurement Information System (PROMIS Global-10) is a valid and reliable patient assessment and consists of ten (10) items that measure physical health, physical functioning, general mental health, emotional distress, satisfaction with social activities and relationships, ability to carry out usual social activities and roles, pain, fatigue and overall quality of life. The response options are presented as 5-point (as well as a single 11-point) rating scales. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score. These scores are then standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient. The PROMIS 10 scores are predictive of healthcare utilization, mortality in general and disease-specific clinical populations.
Visual-Analog Scale (VAS) score | Subject reported outcomes at 3-6 weeks 3-, 6-, 12- and 24-months post-treatment
  This scale has been designed to give subjective pain information as to the degree of knee pain you the patient is currently experiencing. VAS scoring is included in the PROMIS GLOBAL-10 assessment and is not necessary to collect a separate assessment. Applying the VAS, the patient will select a number from 1 (no pain) to 10 (maximum pain) that most closely describes their current pain.
Forgotten Joint Score (FJS-12) | Subject reported outcomes at 3-6 weeks 3-, 6-, 12- and 24-months post-treatment
  The 12 question Forgotten Joint Score (FJS-12) was introduced with the aim of assessing the patients 'joint awareness'. The authors of the score suggest the "higher the score" is more representative of higher-level function after surgery, as to be able to forget about the joint requires the absence of pain and the ability to perform all desired functional tasks without limitation.

CONTACTS AND LOCATIONS:
Overall Officials: Asit Shah, MD, PhD, Study Chair — Chief of Orthopedics - Englewood Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berend KR, Lombardi AV Jr, Mallory TH. Rapid recovery protocol for peri-operative care of total hip and total knee arthroplasty patients. Surg Technol Int. 2004;13:239-47. PMID 15744696
- [Background] Jamsen E, Puolakka T, Eskelinen A, Jantti P, Kalliovalkama J, Nieminen J, Valvanne J. Predictors of mortality following primary hip and knee replacement in the aged. A single-center analysis of 1,998 primary hip and knee replacements for primary osteoarthritis. Acta Orthop. 2013 Feb;84(1):44-53. doi: 10.3109/17453674.2012.752691. Epub 2012 Dec 17. PMID 23244785
- [Background] Durbhakula SR, L. Restoration of Femoral Condylar Anatomy for Achieving Optimum Functional Expectations: Component Design and Early Results. Recon Review 6(3): 5, 2016
- [Background] Durbhakula SD, V.; Durbhakula, N. Restoration of Femoral Condylar Anatomy for Achieving Optimum Functional Expectations: Continuation of an Earlier Study At 5-Year Minimum Follow-Up. Recon Review 9(1): 6, 2019
- [Background] Insall JN, Dorr LD, Scott RD, Scott WN. Rationale of the Knee Society clinical rating system. Clin Orthop Relat Res. 1989 Nov;(248):13-4. PMID 2805470
- [Background] Lyman S, Lee YY, Franklin PD, Li W, Cross MB, Padgett DE. Validation of the KOOS, JR: A Short-form Knee Arthroplasty Outcomes Survey. Clin Orthop Relat Res. 2016 Jun;474(6):1461-71. doi: 10.1007/s11999-016-4719-1. Epub 2016 Feb 29. PMID 26926773
- [Background] Shim J, Hamilton DF. Comparative responsiveness of the PROMIS-10 Global Health and EQ-5D questionnaires in patients undergoing total knee arthroplasty. Bone Joint J. 2019 Jul;101-B(7):832-837. doi: 10.1302/0301-620X.101B7.BJJ-2018-1543.R1. PMID 31256677
- [Background] Thomsen MG, Latifi R, Kallemose T, Barfod KW, Husted H, Troelsen A. Good validity and reliability of the forgotten joint score in evaluating the outcome of total knee arthroplasty. Acta Orthop. 2016 Jun;87(3):280-5. doi: 10.3109/17453674.2016.1156934. Epub 2016 Mar 3. PMID 26937689
- [Background] Boonstra AM, Schiphorst Preuper HR, Reneman MF, Posthumus JB, Stewart RE. Reliability and validity of the visual analogue scale for disability in patients with chronic musculoskeletal pain. Int J Rehabil Res. 2008 Jun;31(2):165-9. doi: 10.1097/MRR.0b013e3282fc0f93. PMID 18467932